CLINICAL TRIAL: NCT00080041
Title: Phase I Trial of Motexafin Gadolinium (MGd) and Docetaxel Administered at 3-Week Intervals for Advanced Solid Tumors
Brief Title: Study of Motexafin Gadolinium and Docetaxel for Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-0214
Record Dates: First submitted 2004-03-22; First posted 2004-03-23 (Estimated); Last update posted 2007-05-15 (Estimated); Status verified 2007-05

CONDITIONS: Breast Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Lung Neoplasms
Keywords: Antineoplastic Combined Chemotherapy Protocols
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Lung Neoplasms | interventions — motexafin gadolinium

INTERVENTIONS:
Drug: Motexafin Gadolinium Injection

SUMMARY:
The primary purpose of this study is to evaluate the safety, toxicities, and dosage for investigational drug Motexafin Gadolinium administered with docetaxel to patients with advanced solid tumors. Secondly, tumor response to the combined treatment will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Histologically or cytologically confirmed diagnosis of cancer (i.e., Unresectable locally advanced or metastatic non-small-cell lung carcinoma (NSCLC) that had progressed during or after one or more chemotherapy regimens; Metastatic breast cancer; Hormone-refractory prostate cancer; Recurrent or refractory ovarian cancer; Sarcoma)
* ECOG performance status score either 0 or 1
* Willing and able to provide written informed consent

Exclusion Criteria:

Laboratory Values of:

* Absolute neutrophil count < 2000/µL
* Platelet count < 100,00/µL
* AST or ALT > 1.5 x the upper limit of normal
* Alkaline phosphatase > 5 x the upper limit of normal
* Bilirubin > ULN
* Creatinine > 2.0 mg/dL

and

* Peripheral neuropathy NCI CTC Grade 3 or higher
* Chemotherapy, radiation therapy, immunotherapy, or systemic biologic
* anticancer therapy within 21 days before beginning study treatment
* Known history of brain metastases or spinal cord compression
* Uncontrolled hypertension
* Myocardial infarction within 6 months before beginning study treatment
* Unstable angina pectoris, uncontrolled congestive heart failure, or uncontrolled serious arrhythmias
* Known sensitivity to or intolerable adverse effects from taxanes or polysorbate 80
* Known history of porphyria (testing not required at screening)
* Known history of glucose-6-phosphate dehydrogenase (G6PD) deficiency (testing not required at screening)
* Known history of HIV infection (testing not required at screening)
* Female who is pregnant or lactating (pregnancy test is required for all female patients of childbearing potential)
* Female of childbearing potential or sexually active male unwilling to use adequate contraceptive protection
* Physical or mental condition that makes patient unable to complete specified follow-up assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20

PRIMARY OUTCOMES:
Determine the Dose Limiting Toxicity at 3 weeks (1 cycle), and the Maximum Tolerated Dose at 24 weeks (6 cycles).

SECONDARY OUTCOMES:
Frequency of tumor responses at weeks 6, 12 and 18.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Cancer Center, Rochester, New York, United States